## THE UNIVERSITY OF BRITISH COLUMBIA



# Division of Urology

## PARTICIPANT INFORMATION AND CONSENT FORM

Title of Study: Effectiveness of Digital Storytelling in Increasing Living Kidney Donor Recruitment in Canada

#### **Principal Investigator:**

**Meghan He, BSc** | Medical Student, Faculty of Medicine, UBC | <a href="mailto:hemeghan@student.ubc.ca">hemeghan@student.ubc.ca</a>, 604 838-1066

## **Co-Investigators:**

**Dr. Christopher Nguan, MD**| Associate Professor, Urologic Sciences, UBC | chris.nguan@ubcurology.com, 604-875-5003

**Dr. Erika Escamilla, MD** | Research Assistant, Urologic Sciences, UBC | <u>tram.nguyen@cw.bc.ca</u>, 604-875-2291

**Dr. David Harriman, MD** | Assistant Professor, Urologic Sciences, UBC | david.harriman@ubcurology.com

## **Background and Study Justification**

In Canada, more than 48,000 patients live with end-stage kidney disease (ESKD) and 29,000 receive weekly dialysis (1). The benefit of kidney transplant, especially a living donor kidney transplant (LDKT), for ESKD patients has been well-established to increase both length and quality of life (2-8). However, the number of solid organ kidney transplants has failed to match the increasing number of ESKD patients in Canada (1). There is thus a large gap between the need for organs and the number of transplants, resulting in 3% of patients dying on the organ waitlist (1).

The need for LDKT is even higher among racialized communities than white patients. Indigenous, East and South Asian, African, Caribbean, and Black communities are 50 to 75 percent less likely to be referred for LDKT, identify donors, complete evaluation, and receive transplant in comparison to white patients in Canada (1). In the United States, African American patients are less likely to receive LDKT than white patients at every transplant center in the country (9). A recent American Society of Transplantation Consensus Conference called for improved transplant education and outreach efforts to target racial barriers to LDKT (10).

Multilevel barriers to LDKT transplant among minority populations have been identified (11). At the individual recipient-donor level, barriers include medical mistrust, low health literacy, religious concerns, and clinical insuitability for donation. At the healthcare provider level, barriers include a lack of cultural competency in transplant education, racially biased perceptions of donation suitability, and limited time for healthcare staff to provide education that addresses racial disparities (12-15). And finally, at the population-community level, there exists a high chronic disease burden among minority populations due to social determinants of health that may reduce the potential donor pool for racialized potential recipients (16-19). Low community awareness about the benefits of and

need for LDKT, low availability of mandated sick leave from work and donor reimbursement further decreases the accessibility of LDKT among racialized populations (20).

Standard of care didactic LKDT education materials have faced numerous health literacy and sociocultural barriers to supporting racialized patients with ESKD (21-23). Namely, no significant change in donation rates resulted from a targeted public education campaign about organ donation in the East Asian communities in British Columbia, Canada (24). This demonstrates the need for culturally appropriate education on kidney transplant that reaches beyond didactic teaching methods.

Storytelling holds the promising potential to close the gap in LDKT access across diverse communities. Recent research has posited that first-person storytelling (FPS) overcomes health literacy and sociocultural barriers to breast cancer, diabetes, hypertension, and smoking cessation interventions (25-31). Several narrative-based transplant education interventions have also proven to be effective in increasing LDKT pursuit among Black patients in America (32-35).

While effective, these education interventions are labour and time intensive and fail to reach the general public and social circles who are not present at the location of transplant education (36). Additionally, the efficacy of interpersonal education interventions has yet to be evaluated in Canadian minority populations, predominantly comprised of South Asian, East Asian and Indigenous communities (37). There is thus a need to analyze the impact of humanities-based LDKT education to narrow the gap in LDKT access in Canada without burdening already limited healthcare resources.

The Living Donation Storytelling Project (LDSP) is an online video library of living donation first-person narratives aiming to inspire more people to consider becoming living donors (36). As of 2020, the library has 118 stories from living donors and kidney recipients sharing their experiences with the challenges, fears, and joys of transplant (36). LDSP is a health-literate and culturally safe approach to LDKT education by virtue of storyteller diversity and its patient-driven approach. The library thus holds the potential to support minority groups in learning about LDKT as a supplement to traditional educational strategies without additional burden for healthcare providers.

### Study Purpose

The purpose of this study is to test the effectiveness of the LDSP as a narrative-based transplant education intervention in encouraging patients with ESKD to pursue LDKT. We will investigate if exposure to the LDSP changes patient readiness and motivation to pursue LDKT to ultimately increase the number of donor inquiries and donor evaluations. We will also test if the LDSP serves as a health-literate and culturally safe education approach that can effectively support racialized communities who have a disproportionately higher need for LDKT.

# Study Objectives

The objectives of this study are to:

- 1: Elucidate if allowing waitlisted transplant patients to watch two videos from the LDSP will increase their readiness and motivation to pursue LDKT.
- 2: Examine if allowing waitlisted transplant patients to watch two videos from the LDSP will increase the number of donor inquiries and donor evaluations.
- 3: Test if the LDSP serves as a health-literate and culturally safe education approach that can effectively support racialized communities in pursuing LDKT.

#### **Outcomes**

| Outcomes | Description | Timeline |
|---|---|---|
| Readiness and | 7 questions assessing stage of change | Baseline + 1-month post- |
| motivation to pursue | 12 questions assessing decisional balance | intervention survey |
| LDKT | | |
| Transplant | 16 questions assessing knowledge about LDKT | |
| Knowledge | | |
| Video Preference | Rate liking after each video | Immediate post- |
| | Rate which of the two videos they preferred | intervention survey |
| Material Accessibility | 1 question assessing ease of understanding | |
| | LDSP stories | |
| Cultural safety | 2 questions assessing LDSP's respect for | |
| | cultural diversity and trustworthiness | |
| Video Impact | 7 questions assessing patient's attitudes | |
| | towards LDSP | |
| Donor Inquiries | Requests for more information about living | 3-month post |
| | donation to the transplant nurse coordinator | intervention EMR review |
| Donor Evaluation | Initiation of the first phase of the clinical | |
| | pathway for living donor evaluation | |

## **Design**

We will conduct a pilot parallel-group, 2-arm randomized control trial comparing the impact of standard LDKT patient education and narratives from the Living Donation Storytelling Project (LDSP) on the attitudes and behaviors of LDKT candidates.

# **Population**

#### **Inclusion Criteria**

- Waitlisted and newly referred kidney transplant candidates at the Vancouver Kidney Transplant Program
- 18 years of age or older

- Able to provide informed consent
- English literate

#### **Exclusion Criteria**

- Inability to understand English and provide informed consent
- Transplant candidates excluded from transplantation based on clinical criteria or other contraindications for transplant
- Unwilling to disclose information on race or ethnicity

#### Recruitment

Study participants will be recruited from Dr. Christopher Nguan and Dr. David Harriman's transplant clinics at Vancouver General Hospital with fully informed consent. Prospective participants will be identified by Dr. Nguan and Dr. Harriman via chart review. A research assistant will describe the study objectives and methods, provide participants with a study information sheet, and ask them if they are interested in participating.

## **Details of Study Procedures**

Participants visiting the transplant clinic at the Vancouver General Hospital will be asked to complete a survey on REDCap following their physician's visit to document their demographics, readiness to pursue transplant, and stage of change in pursuing transplant. Transplant candidates will be randomly assigned to 1 of 2 conditions: (1) a control group that will receive standard-of-care transplant education, and (2) an intervention group that will receive two LDSP videos as a supplement to the standard education.

Participants of the intervention group who self-identified as Caucasian or East Asian on the baseline demographics survey will be shown a series of two videos selected based on race concordance between the viewer (participant) and the storyteller: (1) race non-concordant, (2) race concordant video. Gender will be concordant for all participant-video pairs. The non-concordant video will be shown prior to the concordant video for all participants, and participants will be asked to rate their liking of each video after viewing them one by one. Participants who self-identified as an ethnicity other than Caucasian or East Asian on the baseline demographics survey will be randomly shown two race non-concordant videos. All participants in the intervention arm will also be advised on standard program resources for living donation options.

Patients of the control group will be counseled in standard fashion and connected to recognized resources for living donation options.

A post-intervention surveys will be given via email 1 month after the clinic visit to document their readiness and motivation to pursue LDKT.

3-month post-intervention, we will conduct a chart review to document the number of donor inquiries received and donor evaluations initiated.

## Statistical Analysis

Basic descriptive statistics on participants will be reported as percentages, means, medians and standard deviatiosn. Differences between LDSP versus standard education groups in pre- to postintervention changes in motivation and readiness to pursue LDKT will be examined using linear regression. Results will be summarized as odds ratios and 95% confidence intervals. All analyses will be conducted using R statistical software.

Planned sample size: A convenience sample of 80 patients will be recruited.

#### References

- 1. Canadian Institute for Health Information. <u>Annual statistics on organ replacement in Canada</u>, <u>2012 to 2021</u> [report]. Accessed June 1, 2023.
- 2. de Groot IB, Veen JI, van der Boog PJ, et al. Difference in quality of life, fatigue and societal participation between living and deceased donor kidney transplant recipients. *Clin Transplant*. 2013;27(4):E415-E423.
- 3. Evans RW, Manninen DL, Garrison LP. The quality of life of patients with end-stage renal disease. *New Engl J Med.* 1985;312:553-559
- 4. Molnar MZ, Novak M, Mucsi I. Sleep disorders and quality of life in renal transplant recipients. *Int Urol Nephrol.* 2009;41(2):373-382
- 5. Neipp M, Karavul B, Jackobs S. Quality of life in adult transplant recipients more than 15 years after kidney transplantation. *Transplantation*. 2006;81:1640-1644
- 6. Ortiz F, Aronen P, Koskinen PK. Health-related quality of life after kidney transplantation: who benefits the most. *Transpl Int.* 2014;27(11):1143-1151
- 7. Pinson CW, Feurer ID, Payne JL. Health-related quality of life after different types of solid organ transplantation. *Ann Surg.* 2000;232(4):597-607.
- 8. Network KSC. Alberta annual kidney care report: prevalence of severe kidney disease and use of dialysis and transplantation across Alberta from 2004–2013. Edmonton, AB: Alberta Health Services; 2015.
- 9. Hall EC, James NT, Garonzik Wang JM, et al. Center-level factors and racial disparities in living donor kidney transplantation. *Am J Kidney Dis.* 2012;59(6):849–857. doi:10.1053/j.ajkd.2011.12.021.
- 10. Waterman AD, Morgievich M, Cohen DJ, Butt Z, Chakkera HA, Lindower C, Hays RE, Hiller JM, Lentine KL, Matas AJ, Poggio ED, Rees MA, Rodrigue JR, LaPointe Rudow D; American Society of Transplantation. Living Donor Kidney Transplantation: Improving Education Outside of Transplant Centers about Live Donor Transplantation--Recommendations from a Consensus Conference. Clin J Am Soc Nephrol. 2015 Sep 4;10(9):1659-69. doi: 10.2215/CJN.00950115. Epub 2015 Jun 26. PMID: 26116651; PMCID: PMC4559502.
- 11. Purnell TS, Hall YN, Boulware LE. Understanding and overcoming barriers to living kidney donation among racial and ethnic minorities in the United States. Adv Chronic Kidney Dis. 2012 Jul;19(4):244-51. doi: 10.1053/j.ackd.2012.01.008. PMID: 22732044; PMCID: PMC3385991
- 12. J.Z. Ayanian, P.D. Cleary, J.H. Keogh, S.J. Noonan, J.A. David-Kasdan, A.M. Epstein Physicians' beliefs about racial differences in referral for renal transplantation Am J Kidney Dis, 43 (2004), pp. 350-357
- 13. Ghahramani N. Perceptions of patient suitability for kidney transplantation: a qualitative study comparing rural and urban nephrologists. Paper presented at: American Transplant Conference; May 1-4, 2011; Philadelphia, PA.

- 14. B.L. Kasiske, J.J. Snyder, A.J. Matas, M.D. Ellison, J.S. Gill, A.T. Kausz Preemptive kidney transplantation: the advantage and the advantaged J Am Soc Nephrol, 13 (2002), pp. 1358-1364
- 15. L.E. Boulware, L.A. Meoni, N.E. Fink, *et al.* Preferences, knowledge, communication, and patient-physician discussion of living kidney transplantation in African American families Am J Transplant, 5 (2005), pp. 1503-1512
- 16. B.I. Freedman, B.J. Spray, A.B. Tuttle, V.M. Buckalew The familial risk of end-stage renal disease in African Americans Am J Kidney Dis, 21 (1993), pp. 387-393
- 17. Hajjar, T.A. Kotchen Trends in prevalence, awareness, treatment, and control of hypertension in the United States, 1988–2000 JAMA, 290 (2003), pp. 199-206
- 18. L.E. Barker, K.A. Kirtland, E.W. Gregg, L.S. Geiss, T.J. Thompson Geographic distribution of diagnosed diabetes in the US. A diabetes belt Am J Prev Med, 40 (2011), pp. 434-439
- 19. M. Mujib, Y. Zhang, M.A. Feller, A. Ahmed Evidence of a "heart failure belt" in the Southeastern United States Am J Cardiol, 107 (2011), pp. 935-937
- 20. L.E. Boulware, M.U. Troll, L.C. Plantinga, N.R. Powe The association of state and national legislation with living kidney donation rates in the United States: a National Study Am J Transplant, 8 (2008), pp. 1451-1470
- 21. LaPointe Rudow D, Hays R, Baliga P, Cohen DJ, Cooper M, Danovitch GM, Dew MA, Gordon EJ, Mandelbrot DA, McGuire S, Milton J, Moore DR, Morgievich M, Schold JD, Segev DL, Serur D, Steiner RW, Tan JC, Waterman AD, Zavala EY, Rodrigue JR. Consensus conference on best practices in live kidney donation: recommendations to optimize education, access, and care. Am J Transplant. 2015 Apr;15(4):914-22. doi: 10.1111/ajt.13173. Epub 2015 Feb 3. PMID: 25648884; PMCID: PMC4516059.
- 22. Karavetian M, de Vries N, Elzein H, Rizk R, Bechwaty F. Effect of behavioral stage-based nutrition education on management of osteodystrophy among hemodialysis patients, Lebanon. Patient Educ Couns. 2015 Sep;98(9):1116-22. doi: 10.1016/j.pec.2015.05.005. Epub 2015 May 29. PMID: 26070468.
- 23. Sieverdes JC, Price M, Ruggiero KJ, Baliga PK, Chavin KD, Brunner-Jackson B, Patel S, Treiber FA. Design and approach of the Living Organ Video Educated Donors (LOVED) program to promote living kidney donation in African Americans. Contemp Clin Trials. 2017 Oct;61:55-62. doi: 10.1016/j.cct.2017.07.007. Epub 2017 Jul 5. PMID: 28687348; PMCID: PMC5897101.
- 24. Alsahafi M, Leung L, Partovi N, Yee J, Yoshida EM. Racial differences between solid organ transplant donors and recipients in British Columbia 2005-2009: a follow-up study since the last analysis in 1993-1997. *Transplantation*. 2013;95(11):e70-e71.
- 25. M.W. Kreuter, K. Holmes, K. Alcaraz, B. Kalesan, S. Rath, M. Richert, A. McQueen, N. Caito, L. Robinson, E.M. Clark, Comparing narrative and informational videos to increase mammography in low-income African American women, Patient Educ. Couns. (2010) S6–S14 81 Suppl(Suppl).

- 26. McQueen, M.W. Kreuter, B. Kalesan, K.I. Alcaraz, Understanding narrative effects: the impact of breast cancer survivor stories on message processing, attitudes, and beliefs among African American women, Health Psychol. 30 (6) (2011) 674–682.
- 27. T. Campbell, D. Dunt, J.L. Fitzgerald, I. Gordon, The impact of patient narratives on self-efficacy and self-care in Australians with type 2 diabetes: stage 1 results of a randomized trial, Health Promot. Int. 30 (3) (2015) 438–448.
- 28. B.G. Bokhour, G.M. Fix, H.S. Gordon, J.A. Long, K. DeLaughter, M.B. Orner, C. Pope, T.K. Houston, Can stories influence African-American patients' intentions to change hypertension management behaviors? A randomized control trial, Patient Educ. Couns. 99 (9) (2016) 1482–1488.
- 29. T.K. Houston, J.J. Allison, M. Sussman, W. Horn, C.L. Holt, J. Trobaugh, M. Salas, M. Pisu, Y.L. Cuffee, D. Larkin, S.D. Person, B. Barton, C.I. Kiefe, S. Hullett, Culturally appropriate storytelling to improve blood pressure: a randomized trial, Ann. Internal Med. 154 (2) (2011) 77–84.
- 30. H.L. Nguyen, D.A. Ha, R.J. Goldberg, C.I. Kiefe, G. Chiriboga, H.N. Ly, C.K. Nguyen, N.T. Phan, N.C. Vu, Q.P. Nguyen, J.J. Allison, Culturally adaptive storytelling intervention versus didactic intervention to improve hypertension control in Vietnam- 12 month follow up results: a cluster randomized controlled feasibility trial, PLoS One 13 (12) (2018)e0209912.
- 31. Cherrington, J.H. Williams, P.P. Foster, H.L. Coley, C. Kohler, J.J. Allison, C.I. Kiefe, J.E. Volkman, T.K. Houston, Narratives to enhance smoking cessation interventions among African-American smokers, the ACCE project, BMC Res. Notes 8 (2015) 567.
- 32. Weng, Francis L. MD, MSCE1,2; Davis, LaShara A. PhD1,3; Ohman-Strickland, Pamela A. PhD2; Waterman, Amy D. PhD4,5. Destination Transplant: Protocol for a Parallel-group Randomized Trial of an Educational Intervention to Increase Kidney Transplant Among Black People on the Transplant Waiting List. Transplantation Direct 7(4):p e683, April 2021. | DOI: 10.1097/TXD.00000000001136
- 33. Waterman AD, Peipert JD. An Explore Transplant Group Randomized Controlled Education Trial to Increase Dialysis Patients' Decision-Making and Pursuit of Transplantation. Prog Transplant. 2018 Jun;28(2):174-183. doi: 10.1177/1526924818765815. Epub 2018 Apr 26. PMID: 29699451.
- 34. Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, Falcone B, Ephraim PL, Jaar BG, Gimenez L, Choi M, Senga M, Kolotos M, Lewis-Boyer L, Cook C, Light L, DePasquale N, Noletto T, Powe NR. Effectiveness of educational and social worker interventions to activate patients' discussion and pursuit of preemptive living donor kidney transplantation: a randomized controlled trial. Am J Kidney Dis. 2013 Mar;61(3):476-86. doi: 10.1053/j.ajkd.2012.08.039. Epub 2012 Oct 22. PMID: 23089512; PMCID: PMC3710736.
- 35. Rodrigue JR, Cornell DL, Lin JK, Kaplan B, Howard RJ. Increasing live donor kidney transplantation: a randomized controlled trial of a home-based educational intervention. Am J Transplant. 2007 Feb;7(2):394-401. doi: 10.1111/j.1600-6143.2006.01623.x. Epub 2006 Dec 6. PMID: 17173659.

- 36. Waterman AD, Wood EH, Ranasinghe ON, Faye Lipsey A, Anderson C, Balliet W, Holland-Carter L, Maurer S, Aurora Posadas Salas M. A Digital Library for Increasing Awareness About Living Donor Kidney Transplants: Formative Study. JMIR Form Res. 2020 Jul 21;4(7):e17441. doi: 10.2196/17441. PMID: 32480362; PMCID: PMC7404010.
- 37. Statistics Canada. Immigration and ethnocultural diversity: key results from the 2016 Census. https://www150.statcan.gc.ca/n1/daily-quotidien/171025/dq171025b-info-eng.htm. Published 2017. Accessed February 10, 2021.